CLINICAL TRIAL: NCT04519879
Title: A Randomized Phase 2 Trial of White Button Mushroom Supplement in Patients With Biochemically Recurrent Prostate Cancer Following Local Therapy and in Therapy Na?ve Patients With Favorable Risk Prostate Cancer Undergoing Active Surveillance
Brief Title: White Button Mushroom Sup for the Reduction of PSA in Pts With Biochemically Rec or Therapy Naive Fav Risk Prostate CA
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 19296; NCI-2019-05587 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 19296 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2019-09-12; First posted 2020-08-20 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Prostate Adenocarcinoma; PSA Failure; PSA Progression; Recurrent Prostate Carcinoma; Stage I Prostate Cancer AJCC v8; Stage IIA Prostate Cancer AJCC v8; Stage IIB Prostate Cancer AJCC v8; Stage IIC Prostate Cancer AJCC v8; Stage IIIA Prostate Cancer AJCC v8; Stage IIIC Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Watchful Waiting; Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm IA (white mushroom extract) (Experimental): Patients receive white button mushroom extract PO BID on day 1. Treatment repeats every 4 weeks for cycles 1-3 then every 12 weeks for cycles 4-6 (36 weeks) in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Questionnaire Administration; Drug: White Button Mushroom Extract
- Arm IB (clinical observation) (Active Comparator): Patients undergo clinical observation for 12 weeks. If PSA continues to increase, patients have the option to receive the white button mushroom extract as in arm IA.
  Interventions: Other: Clinical Observation; Other: Questionnaire Administration
- Arm IIA (white mushroom extract) (Experimental): Patients receive white mushroom extract PO BID on day 1. Treatment repeats every 12 weeks for 4 cycles (48 weeks) in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Questionnaire Administration; Drug: White Button Mushroom Extract
- Arm IIB (active surveillance) (Active Comparator): Patients undergo active surveillance for 48 weeks.
  Interventions: Other: Patient Observation; Other: Questionnaire Administration

INTERVENTIONS:
Other: Clinical Observation — Undergo clinical observation
  Other Names: observation
  Arms: Arm IB (clinical observation)
Other: Patient Observation — Undergo active surveillance
  Other Names: Active Surveillance; deferred therapy; expectant management; observation; Watchful Waiting
  Arms: Arm IIB (active surveillance)
Other: Questionnaire Administration — Ancillary studies
Drug: White Button Mushroom Extract — Given PO
  Other Names: WBM Extract
  Arms: Arm IA (white mushroom extract); Arm IIA (white mushroom extract)

SUMMARY:
This phase II trial studies how well white button mushroom supplement works in reducing prostate-specific antigen (PSA) levels in patients with prostate cancer that has come back (recurrent) or has favorable risk and has not undergone any therapy (therapy naive). PSA is a blood marker of prostate growth. White button mushroom supplement may affect PSA level, various parameters of immune system and levels of hormones that may have a role in prostate cancer growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the proportion of patients with any prostate specific antigen (PSA) reduction at 12 weeks (~3 months) in observation + white button mushroom (WBM) supplement arm and observation only arm (control arm). (Cohort 1) II. To assess relative change in PSA at 48 weeks (~12 months) from baseline with or without WBM treatment. (Cohort 2)

SECONDARY OBJECTIVES:

I. To evaluate, adverse events, PSA-response rate and time to PSA progression. (Cohort 1) II. To evaluate adverse events, time to initiation of additional therapy and progression. (Cohort 2)

EXPLORATORY OBJECTIVES:

I. To characterize the immunomodulatory effects of WBM supplement in serial blood samples. (Cohort 1) II. To assess the effect of therapy with WBM on sexual function. (Cohort 1) III. To assess the effect of WBM on Gleason grade in prostate cancer subjects on active surveillance. (Cohort 2) IV. To characterize the immunomodulatory effects of WBM supplement in serial blood samples and in tumor tissue. (Cohort 2) V. To characterize changes in cancer signaling pathways in tumor tissue after intake of WBM supplement. (Cohort 2) VI. To assess the effect of WBM supplement on sexual function. (Cohort 2)

OUTLINE: Patients are assigned to 1 of 2 cohorts.

COHORT I: Biochemically recurrent prostate cancer patients are randomized to 1 of 2 arms.

ARM IA: Patients receive white button mushroom extract orally (PO) twice daily (BID) on day 1. Treatment repeats every 4 weeks for cycles 1-3 then every 12 weeks for cycles 4-6 (36 weeks) in the absence of disease progression or unacceptable toxicity.

ARM IB: Patients undergo clinical observation for 12 weeks. If PSA continues to increase, patients have the option to receive the white button mushroom extract as in arm IA.

COHORT II: Therapy naive favorable risk prostate cancer patients are randomized to 1 of 2 arms.

ARM IIA: Patients receive white mushroom extract PO BID on day 1. Treatment repeats every 12 weeks for 4 cycles (48 weeks) in the absence of disease progression or unacceptable toxicity.

ARM IIB: Patients undergo active surveillance for 48 weeks.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative
* For therapy naive favorable risk prostate cancer (cohort 2 only): agreement to undergo baseline and 48 week prostate biopsy
* Willing to forego non-study supplements containing mushroom for the duration of the study
* Eastern Cooperative Oncology Group (ECOG) =< 2
* Histologically or cytologically confirmed history of adenocarcinoma of the prostate
* BIOCHEMICALLY RECURRENT PROSTATE CANCER COHORT (COHORT 1) ONLY: PSA failure defined as:

  * PSA of >= 0.2 ng/mL that has increased above nadir following prostatectomy, OR
  * PSA increase of 2.0 ng/mL above post-therapy nadir if other primary local therapy was used instead of prostatectomy
  * NOTE: PSA value must be increasing based on 2 consecutive measurements taken at least 2 weeks apart
* BIOCHEMICALLY RECURRENT PROSTATE CANCER COHORT (COHORT 1) ONLY: Testosterone levels > 50 ng/dL
* BIOCHEMICALLY RECURRENT PROSTATE CANCER COHORT (COHORT 1) ONLY: Received any number of primary local therapies, defined as:

  * Radical prostatectomy
  * External beam radiation therapy
  * Radioactive seed implantation
  * Cryotherapy
  * High-intensity focused ultrasound (HIFU)
* BIOCHEMICALLY RECURRENT PROSTATE CANCER COHORT (COHORT 1) ONLY: May have received up to 24 months of neoadjuvant/adjuvant androgen deprivation therapy in conjunction with primary local therapy. Androgen deprivation therapy must have been completed > 6 months from day (D)1 of the study
* BIOCHEMICALLY RECURRENT PROSTATE CANCER COHORT (COHORT 1) ONLY: Neoadjuvant/adjuvant cytotoxic chemotherapy must have been completed > 6 months from day (D)1 of the study
* BIOCHEMICALLY RECURRENT PROSTATE CANCER COHORT (COHORT 1) ONLY: No clinical or radiographic evidence of metastatic disease within 2 months prior to day 1 of protocol therapy. If metastatic disease is detected by positron emission tomography (PET) imaging only patients are eligible as long as no metastatic disease is noted on computed tomography (CT) scan (or magnetic resonance imaging [MRI]) and bone scan
* THERAPY NAIVE FAVORABLE RISK PROSTATE CANCER COHORT (COHORT 2) ONLY: Adenocarcinoma of the prostate diagnosed =< 12 months of protocol screening and has elected active surveillance as preferred management plan OR already on active surveillance
* THERAPY NAIVE FAVORABLE RISK PROSTATE CANCER COHORT (COHORT 2) ONLY: Clinical stage T1c-T2a as defined below:

  * T1c: Tumor identified by needle biopsy found in one or both sides, but not palpable
  * T2a: Tumor involves one-half of one side or less
* THERAPY NAIVE FAVORABLE RISK PROSTATE CANCER COHORT (COHORT 2) ONLY: Gleason score =< 6 (grade group 1) or Gleason 3+4 (grade group 2)
* THERAPY NAIVE FAVORABLE RISK PROSTATE CANCER COHORT (COHORT 2) ONLY: Adequate biopsy of at least 10 biopsy cores
* THERAPY NAIVE FAVORABLE RISK PROSTATE CANCER COHORT (COHORT 2) ONLY: No prior therapy for prostate cancer defined as:

  * Local therapy including surgery , radiation or focal therapy (cryoablation, HIFU, light)
  * Systemic therapy (hormonal, immunotherapy, targeted, chemotherapy). Subjects who have used 5-alpha reductase inhibitor (e.g. finasteride or dutasteride) > 6 months prior to D1 of protocol therapy will be allowed
* Platelets > 100,000 /mm^3 (within 28 days prior to day 1 of protocol therapy)
* Hemoglobin > 8 g/dL (within 28 days prior to day 1 of protocol therapy)
* Aspartate aminotransferase, alanine aminotransferase, < 3 x upper limit of normal (ULN) (within 28 days prior to day 1 of protocol therapy)
* Total bilirubin < 2 x ULN (within 28 days prior to day 1 of protocol therapy)
* Creatinine < 2 x ULN (within 28 days prior to day 1 of protocol therapy)

Exclusion Criteria:

* Other concomitant investigational anti-cancer therapy/ vaccines/biologics, corticosteroids with > 10 mg of prednisone equivalent dose
* Therapy with mushroom supplements within last 3 months of randomization
* BIOCHEMICALLY RECURRENT PROSTATE CANCER COHORT (COHORT 1) ONLY: Neoadjuvant/adjuvant androgen derivation therapy lasting > 24 months or within 6 months prior to day 1 of protocol therapy
* BIOCHEMICALLY RECURRENT PROSTATE CANCER COHORT (COHORT 1) ONLY: Neoadjuvant/adjuvant chemotherapy within 6 months prior to day 1 of protocol therapy
* BIOCHEMICALLY RECURRENT PROSTATE CANCER COHORT (COHORT 1) ONLY: Prior therapy for recurrent prostate cancer (unless given as a component of attempted curative salvage treatment including salvage radiation therapy, and completed > 6 months before day 1 of protocol therapy):

  * Chemotherapy
  * Androgen deprivation therapy
  * Immunotherapy
  * Targeted therapy
* Known history of allergic reaction to mushrooms
* Clinically significant uncontrolled illness
* Active infection requiring treatment
* Uncontrolled congestive heart failure, cardiac arrhythmia
* History of other primary non-skin malignancy within previous 2 years unless treated with curative intent and in remission
* Any other condition that would, in the Investigator?s judgment, contraindicate the patient?s participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2026-05-14 (Estimated); Study Completion 2026-05-14 (Estimated)

PRIMARY OUTCOMES:
Prostate-specific antigen (PSA) (ng/mL) levels (Cohort 1) | At 12 weeks
  For continuous variables, descriptive statistics (number [n], mean, standard deviation, standard error, median range) will be provided. For categorical variables, patient counts and percentages will be provided.
Relative change in PSA (Cohort 2) | Baseline up to 48 weeks
  The relative difference in PSA will be measured as log (48 week PSA/baseline PSA). Undetectable PSA at 48 weeks will be coded as the low end of the lab measurement range for PSA. This measure of relative difference will be compared between the white button supplement (WBM) + active surveillance and active surveillance only patients. For continuous variables, descriptive statistics (n, mean, standard deviation, standard error, median range) will be provided. For categorical variables, patient counts and percentages will be provided.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 48 weeks
  Will be defined per National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0. Grade 2 serious adverse events and all grade 3-5 adverse events will be reported in the e-case report forms. Observed toxicities will be summarized in terms of type (organ affected or laboratory determination), severity, attribution, time of onset, probable association with the study treatment and reversibility or outcome.
Proportion of patients with PSA response (Cohort 1) | Up to 48 weeks
  Will be defined as the sum of complete (PSA-normalization) and partial responders (PSA-partial response) vs non-responders. For continuous variables, descriptive statistics (number [n], mean, standard deviation, standard error, median range) will be provided. For categorical variables, patient counts and percentages will be provided.
Time to PSA progression (Cohort 1) | Time from randomization to PSA progression, assessed up to 48 weeks
  For continuous variables, descriptive statistics (number [n], mean, standard deviation, standard error, median range) will be provided. For categorical variables, patient counts and percentages will be provided.
Time to initiation of additional therapy (Cohort 2) | Baseline up to 48 weeks
  For continuous variables, descriptive statistics (n, mean, standard deviation, standard error, median range) will be provided. For categorical variables, patient counts and percentages will be provided.
Time to progression (Cohort 2) | From randomization to progression, assessed up to 48 weeks
  Will be defined as any Gleason grade 4 or 5 upon repeat biopsy or conversion from 3+4 to 4+3 or higher, prostate cancer is found in a greater number of prostate biopsy cores, prostate cancer occupies a greater extent of the prostate biopsy cores, PSA > 100 ng/mL. For continuous variables, descriptive statistics (n, mean, standard deviation, standard error, median range) will be provided. For categorical variables, patient counts and percentages will be provided.

OTHER OUTCOMES:
Change in temporal levels of circulating myeloid-derived suppressor cells (MDSCs) | Baseline to 48 weeks
  Will be studies within the peripheral blood mononuclear cell (PBMC) compartment. Will evaluate the relative change in prostate cancer-associated MDSCs after 12 weeks of WBM supplement intake in borderline resectable pancreatic cancer patients versus in those on observation using a two group t-test. Results for cohort 1 will be confirmed by analyzing prostate cancer-associated MDSCs in cohort 2 as well (change from baseline to 48 weeks).
Change in temporal levels of pro-/anti-inflammatory mediators | Baseline up to 48 weeks
  Will include cytokines/growth factors/chemokines, including IL-15 in plasma. Will evaluate the baseline correlatives and the relative role of treatment in a multivariate exploratory analysis.
Sexual function | Up to 48 weeks
  Will be evaluated by the sexual function questionnaire, including the Sexual Health Inventory for Men score. The Sexual Health Inventory for Men (SHIM) Questionnaire scoring system will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Clayton S Lau, Principal Investigator — City of Hope Medical Center
Locations (7):
- United States (7):
  - City of Hope Medical Center, Duarte, California
  - City of Hope at Glendora, Glendora, California
  - City of Hope at Irvine Lennar, Irvine, California
  - City of Hope Rancho Cucamonga, Rancho Cucamonga, California
  - John Wayne Cancer Institute, Santa Monica, California
  - City of Hope South Pasadena, South Pasadena, California
  - City of Hope West Covina, West Covina, California

REFERENCES:
- [Derived] Wang X, Ma S, Twardowski P, Lau C, Chan YS, Wong K, Xiao S, Wang J, Wu X, Frankel P, Wilson TG, Synold TW, Presant C, Dorff T, Yu J, Sadava D, Chen S. Reduction of myeloid-derived suppressor cells in prostate cancer murine models and patients following white button mushroom treatment. Clin Transl Med. 2024 Oct;14(10):e70048. doi: 10.1002/ctm2.70048. PMID 39390760